CLINICAL TRIAL: NCT03493698
Title: A Phase 1, Open-label, Fixed-Sequence, Drug-Drug Interaction Study Between Multiple Oral Doses of Inarigivir Soproxil and a Single Oral Dose of Midazolam in Healthy Subjects
Brief Title: A Fixed-Sequence, Drug-Drug Interaction Study Between Multiple Oral Doses of Inarigivir Soproxil and a Single Oral Dose of Midazolam in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: F-star Therapeutics, Inc. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SBP-9200-HBV-202; 2018-000607-16 (EudraCT Number)
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Drug Interaction Potentiation
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A: Midazolam (Experimental): All subjects will receive a single oral dose of 2 mg Midazolam on Day 1
  Interventions: Drug: Midazolam
- Treatment B and C: Inarigivir (Experimental): All subjects will receive a single oral dose of 400 mg Inarigivir on Day 3, Day 6-18
  Interventions: Drug: Inarigivir
- Treatment D: Inarigivir with Midazolam (Experimental): All subjects will receive a single oral dose of 400 mg Inarigivir coa administered with a single oral dose of 2 mg Midazolam on Day 19
  Interventions: Drug: Midazolam; Drug: Inarigivir

INTERVENTIONS:
Drug: Midazolam — Midazolam
  Arms: Treatment A: Midazolam; Treatment D: Inarigivir with Midazolam
Drug: Inarigivir — Inarigivir
  Other Names: Inarigivir Soproxil, SB 9200
  Arms: Treatment B and C: Inarigivir; Treatment D: Inarigivir with Midazolam

SUMMARY:
This is a single center, open-label, fixed sequence study to investigate the effect of multiple oral dosing of Inarigivir Soproxil and a single oral dose of Midazolam in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Gender : male or female
2. Age : 18-55 years, inclusive, at screening
3. Body mass index (BMI) : 18.0-30.0 kg/m2, inclusive, at screening
4. Status : healthy subjects
5. At screening, females must be non-pregnant and non-lactating, or of non-childbearing potential (either surgically sterilized or physiologically incapable of becoming pregnant, or at least 1 year post-menopausal [amenorrhoea duration of 12 consecutive months]); non-pregnancy will be confirmed for all females by a serum pregnancy test conducted at screening, and a urine pregnancy test at each admission and at follow-up
6. Female subjects of childbearing potential, with a fertile male sexual partner, must agree to use adequate contraception from screening until 90 days after the follow-up visit. Adequate contraception is defined as using a non-hormonal intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm or cervical cap, or a condom; please note that hormonal contraceptives are not allowed. Also, total abstinence, in accordance with the lifestyle of the subject, is acceptable
7. Male subjects, if not surgically sterilized, must agree to use adequate contraception and not donate sperm from admission to the clinical research center until 90 days after the follow-up visit. Adequate contraception for the male subject (and his female partner) is defined as using hormonal contraceptives or an intrauterine device, combined with at least 1 of the following forms of contraception: a diaphragm or cervical cap, or a condom. Also, total abstinence, in accordance with the lifestyle of the subject is acceptable
8. All prescribed medication, including hormonal contraceptives for female subjects, must have been stopped at least 30 days prior to admission to the clinical research center
9. All over-the-counter medication, vitamin preparations and other food supplements, or herbal medications (eg, St. John's Wort) must have been stopped at least 14 days prior to admission to the clinical research center. An exception is made for paracetamol, which is allowed up to admission to the clinical research center
10. Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, energy drinks) and grapefruit (juice) from 72 hours prior to admission to the clinical research center
11. Good physical and mental health on the basis of medical history, physical examination, clinical laboratory, electrocardiogram (ECG) and vital signs, as judged by the PI
12. Willing and able to sign the ICF

Exclusion Criteria:

1. Employee of PRA or the Sponsor
2. History of relevant drug and/or food allergies
3. Using tobacco products within 60 days prior to the first drug administration
4. History of alcohol abuse or drug addiction (including soft drugs like cannabis products)
5. Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants and alcohol) at screening and admission to the clinical research center
6. Average intake of more than 24 units of alcohol per week (1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
7. Positive screen for hepatitis B surface antigen (HBsAg), anti-HCV antibodies or anti-human immunodeficiency virus (HIV) 1 and 2 antibodies
8. Participation in a drug study within 60 days prior to the first drug administration in the current study. Participation in more than 4 other drug studies in the 12 months prior to the first drug administration in the current study
9. Donation or loss of more than 100 mL of blood within 60 days prior to the first drug administration. Donation or loss of more than 1.5 liters of blood (for male subjects) / more than 1.0 liters of blood (for female subjects) in the 10 months prior to the first drug administration in the current study
10. Significant and/or acute illness within 5 days prior to the first drug administration that may impact safety assessments, in the opinion of the PI

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen van de Wetering, Principal Investigator — PRA Health Sciences
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each subject was expected to complete treatment groups A, B, C and D; sequentially.
Groups:
- Sequential Single, Multi-day & Combo Midazolam and Inarigivir: A: All subjects will receive a single oral dose of 2 mg Midazolam on Day 1
  B: All subjects will receive a single oral dose of 400 mg Inarigivir on Day 3
  C: All subjects receive oral dose of 400 mg Inarigivir once daily from Day 6 to Day 18
  D: All subjects will receive a single oral dose of 400 mg Inarigivir coadministered with a single oral dose of 2 mg Midazolam on Day 19
Period: Treatment Period A
Arm/Group | Sequential Single, Multi-day & Combo Midazolam and Inarigivir
Started | 17
Completed | 17
Not Completed | 0
Period: Treatment Period B
Arm/Group | Sequential Single, Multi-day & Combo Midazolam and Inarigivir
Started | 17
Completed | 17
Not Completed | 0
Period: Treatment Period C
Arm/Group | Sequential Single, Multi-day & Combo Midazolam and Inarigivir
Started | 17
Completed (One subject withdrawn from the study on Day 9 and was replaced) | 15
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: Treatment Period D
Arm/Group | Sequential Single, Multi-day & Combo Midazolam and Inarigivir
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sequential Single, Multi-day & Combo Midazolam and Inarigivir
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age was 30 years; Individual age ranged between 18 and 46 years
  years | 30 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 17
BMI [Mean (Standard Deviation); unit: kg/m^2] — Individual BMI ranged between 19.3 and 30.0 kg/m2
  kg/m^2 | 25.5 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Steady-state Oral Inarigivir on the Single Dose Pharmacokinetics (PK) of Oral Midazolam in Healthy Subjects (Cmax)
Description: Comparison of Cmax for midazolam between Treatments A and D.
Time Frame: Day 1 Treatment A and Day 19 Treatment D, respectively
Population: All subjects who received at least one dose of midazolam and had sufficient concentration-time data to reliably estimate PK parameters
Measure: Mean (Full Range); unit: ng/mL
Groups:
- Treatment B and C: Inarigivir: B: All subjects will receive a single oral dose of 400 mg Inarigivir on Day 3
  C: All subjects receive oral dose of 400 mg Inarigivir once daily from Day 6 to Day 18
  Inarigivir: Inarigivir
- Treatment D: Inarigivir With Midazolam: All subjects will receive a single oral dose of 400 mg Inarigivir coadministered with a single oral dose of 2 mg Midazolam on Day 19
  Midazolam: Midazolam
  Inarigivir: Inarigivir
Arm/Group | Treatment A: Midazolam | Treatment B and C: Inarigivir | Treatment D: Inarigivir With Midazolam
Number analyzed (Participants) | 17 | 0 | 15
ng/mL | 12.4 [6.19 to 21.4] |  | 13.0 [7.54 to 21.0]

2. Primary Outcome: Effect of Steady-state Oral Inarigivir on the Single Dose Pharmacokinetics (PK) of Oral Midazolam in Healthy Subjects (AUC0-t)
Description: Comparison of AUC0-t for midazolam between Treatments A and D.
Time Frame: Day 1 Treatment A and Day 19 Treatment D, respectively
Population: This outcome measure was prespecified for treatment groups A and D only.
Measure: Mean (Full Range); unit: h.ng/ml
Arm/Group | Treatment A: Midazolam | Treatment B and C: Inarigivir | Treatment D: Inarigivir With Midazolam
Number analyzed (Participants) | 17 | 0 | 15
h.ng/ml | 29.9 [16.2 to 57.7] |  | 28.7 [15.6 to 44.6]

3. Primary Outcome: Effect of Steady-state Oral Inarigivir on the Single Dose Pharmacokinetics (PK) of Oral Midazolam in Healthy Subjects (AUC0-inf )
Description: Comparison of AUC0-inf for midazolam between Treatments A and D.
Time Frame: Day 1 Treatment A and Day 19 Treatment D, respectively
Population: This outcome measure was prespecified for treatment groups A and D only.
Measure: Mean (Full Range); unit: h.ng/ml
Arm/Group | Treatment A: Midazolam | Treatment B and C: Inarigivir | Treatment D: Inarigivir With Midazolam
Number analyzed (Participants) | 17 | 0 | 15
h.ng/ml | 31.5 [16.7 to 61.6] |  | 30.5 [16.6 to 49.4]

4. Secondary Outcome: Number of Participants With Clinical Relevant Clinical Laboratory, Vital Signs, 12-lead ECG, or Physical Examination
Description: Safety and tolerability were measured via clinical laboratory evaluations, vital signs, 12-lead ECG, or physical examination
Time Frame: Day -1 to Day 20 and Follow-up (5-9 days post-treatment)
Population: All participants analyzed
Measure: Count of Participants; unit: Participants
Groups:
- Treatment B: Inarigivir: B: All subjects will receive a single oral dose of 400 mg Inarigivir on Day 3
  Inarigivir: Inarigivir
- Treatment C: Inarigivir: C: All subjects receive oral dose of 400 mg Inarigivir once daily from Day 6 to Day 18
  Inarigivir: Inarigivir
Arm/Group | Treatment A: Midazolam | Treatment B: Inarigivir | Treatment C: Inarigivir | Treatment D: Inarigivir With Midazolam
Number analyzed (Participants) | 17 | 15 | 15 | 15
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: PK of Inarigivir After Single and Multiple Oral Doses in Healthy Subjects (AUC)
Description: A summary of the main plasma PK parameters for inarigivir, Rp-SB 9000, Sp-SB 9000, and Rp-SB 9000 and Sp-SB 9000 combined after a single oral dose of 400 mg inarigivir on Day 3 (Treatment B) and after the last of 14 consecutive daily oral doses of 400 mg inarigivir from Day 6 to 19 (Treatment D)
Time Frame: Day 3 and Day 6 to 19
Population: All subjects in treatment arms B and D who received inarigivir and had sufficient concentration-time data to reliably estimate PK parameters
Measure: Mean (Full Range); unit: h.ng/ml
Arm/Group | Treatment B: Inarigivir | Treatment D: Inarigivir With Midazolam
Number analyzed (Participants) | 17 | 15
h.ng/ml
  Day 3 AUC0-t (h.ng/mL): number analyzed (Participants) | 17 | 0
  Day 3 AUC0-t (h.ng/mL) | 0.914 [0.129 to 3.23] |
  Day 3AUC0-inf (h.ng/mL): number analyzed (Participants) | 9 | 0
  Day 3AUC0-inf (h.ng/mL) | 1.19 [0.609 to 2.44] |
  Day 19 AUC0-t (h.ng/mL): number analyzed (Participants) | 0 | 15
  Day 19 AUC0-t (h.ng/mL) |  | 0.951 [0.238 to 2.26]

6. Secondary Outcome: PK of Inarigivir After Single and Multiple Oral Doses in Healthy Subjects (Cmax)
Description: as for outcome 5
Time Frame: Day 3 and Day 6 to 19
Population: as for outcome 5
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Treatment B: Inarigivir | Treatment D: Inarigivir With Midazolam
Number analyzed (Participants) | 17 | 15
ng/mL | 0.886 [0.182 to 2.77] | 0.991 [0.221 to 4.07]

ADVERSE EVENTS:
Time Frame: 20 days
Arm/Group | Treatment A: Midazolam | Treatment B: Inarigivir | Treatment C: Inarigivir | Treatment D: Inarigivir With Midazolam
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 4/17 | 4/17 | 7/17 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: Midazolam (N=17) | Treatment B: Inarigivir (N=17) | Treatment C: Inarigivir (N=17) | Treatment D: Inarigivir With Midazolam (N=15)
Fatigue (General disorders) | 1 | 2 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 1 | 0
Sensation of Foreign Body (General disorders) | 0 | 0 | 1 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Laryngeal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 (2) | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Affect Lability (Psychiatric disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT03493698/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT03493698/SAP_001.pdf